CLINICAL TRIAL: NCT07175077
Title: 7T Brain MRI Scan for Micro-brain Metastasis (microBM) Detection for Patients With Small-cell Lung Cancer (SCLC), Who Decline Prophylactic Cranial Irradiation (PCI)
Status: Recruiting | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Principal Investigator, Bo Lu, CHAIR & PROFESSOR, DEPARTMENT OF RADIATION ONCOLOGY, University of Missouri-Columbia
Other Study IDs: 2122797
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Small-cell Lung Cancer; Brain Metastases
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: 7t MRI — 7t brain MRI followed by up to 12 months of standard of care 1.5t/3t MRI scans

SUMMARY:
Comparison of a 7t MRI to standard of care 1.5t/3t MRI scans to determine if earlier detection of brain metastases are possible on a 7t.

DETAILED DESCRIPTION:
This study is looking at patients diagnosed with small-cell lung cancer & have declined prophylactic cranial irradiation. Patients must have had a 1.5t/3t MRI performed within 4 weeks of consenting to the trial that was negative for brain metastases. Patients will then undergo a 7t MRI & be followed for their standard of care scans for 12 months or until confirmed metastases are detected. Once a patient has confirmed brain mets, their standard of care scans will be used for an analysis compared to the 7t scan to determine if earlier detection of brain micro metastases are feasible.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically confirmed diagnosis of small-cell lung cancer (SCLC). • Patient must have an MRI of the brain, performed within 4 weeks prior to consent, documenting no evidence of brain metastases or leptomeningeal disease.
* Patient also must not have a history of brain metastases or leptomeningeal disease.
* Patient must refuse PCI and agree to surveillance with brain MRI scans (1.5T/3T).
* Patient must be ≥ 18 years of age.
* Patient must have ECOG Performance Status of 0-2
* Patients must be able to tolerate the 7T MRI

Exclusion Criteria:

* Patient must not have a contraindication to an MRI, such as implanted metal devices or foreign bodies.
* Patient must not have a contraindication to gadolinium contrast administration during MR imaging.
* Patient must not have other metastatic malignancies requiring current active treatment.
* Pregnant patients are excluded. Pregnancy status will be confirmed verbally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to clinic & who have declined PCI will be presented and offered the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
7t MRI Brain Metastases Detection | 3, 6, 9, 12 months after 7T MRI
  Comparison of 7t MRI to 1.5t/3t to determine if the 7t MRI was able to detect metastases prior to a 1.5t/3t MRI

CONTACTS AND LOCATIONS:
Overall Officials: Bo Lu, MD, Principal Investigator — CHAIR & PROFESSOR, DEPARTMENT OF RADIATION ONCOLOGY
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No